CLINICAL TRIAL: NCT03021564
Title: Prospective Multi-centre Observational Study on the Epidemiology, Risk Factors and Consequences of Unexpected Cardiac Arrest in Intensive Care Units.
Brief Title: Unexpected Cardiac Arrest in Intensive Care Unit
Acronym: ACIR
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/P04/049
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cardiopulmonary resuscitation — Basic cardiopulmonary resuscitation : external electric shock, external cardiac massage, adrenaline injection ...

SUMMARY:
Unexpected cardiac arrest involves approximately 0.5 to 5% of patients admitted in Intensive Care Unit (ICU). Even if they have a technical environment conducive to prompt diagnosis and prompt treatment, patients hospitalized in ICU suffer from chronic illnesses and organ failure(s) that obscure the prognosis of cardiac arrest. Although extra cardiac arrhythmias or intra-hospital arrests are the subject of numerous publications, few studies specifically focus on unexpected cardiac arrest in ICU (none in France). The objective of our work is to produce a prospective epidemiological description of unexpected cardiac arrest in in French ICUs.

DETAILED DESCRIPTION:
Unexpected cardiac arrest in ICU corresponds to cardiovascular arrest leading to at least one cardiopulmonary resuscitation technique (external cardiac massage and / or electric shock). They account for about 0.5 to 5% of admissions to intensive care units. Even if they benefit from a technical environment conducive to prompt diagnosis and rapid management, Resuscitated patients suffer from chronic diseases and organ failure (s) that darken the prognosis. Etiologies of unexpected cardiac arrest in ICU are rarely described in the literature. Their specificity comes from the fact that they can be related to patient's medical characteristics, but also to deleterious effects of supportive techniques in place at the time of circulatory arrest (respiratory assistance, vasopressor drugs, extracorporeal circulation ...). These same techniques may also reduce the effectiveness of cardiopulmonary resuscitation (cardiorespiratory interactions of respiratory assistance, pro-arrhythmogenic effect of vasopressor drugs, haemodynamic repercussion of extracorporeal circulation). Although cardiac arrests have been published extensively out of or in-hospital, there are few studies specifically concerning unexpected cardiac arrest in ICU (none in France). The prognosis is different: after an unexpected cardiac arrest in ICU, 50% of the patients recover a spontaneous cardiac activity but only 15% leave alive from the hospital (3 to 4% with a good functional autonomy). A prospective description of risk factors, circumstances and consequences in the medium term would identify (and prevent) risky situations and identify, among those at risk for unexpected cardiac arrest, those for whom a cardiopulmonary resuscitation is justified.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unexpected cardiac arrest during his / her hospitalization in the ICU
* Patients who have benefited from at least one basic cardiopulmonary resuscitation technique by the ICU team to treat this circulatory arrest (external electric shock, external cardiac massage, adrenaline injection ...)
* Patients with multiple unexpected cardiac arrest during hospitalization will be included only for the first circulatory arrest.

Exclusion Criteria:

* Patients with unexpected cardiac that have not been resuscitated.
* Patients in cardiac arrest at admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in intensive care unit during the study period and presenting an unexpected cardiac arrest will be included
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Leloup, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (45):
- France (45):
  - CH Agen, Agen
  - CHU Angers, Angers
  - CH Angouleme, Angoulême
  - CH Angoulême, Angoulême
  - CH Arras, Arras
  - GH Carnelle Portes de l'Oise, Beaumont
  - CH Béthune, Béthune
  - CH Blois, Blois
  - APHP, Bobigny
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CH Cahors, Cahors
  - CH Chartres, Chartres
  - CH Cholet, Cholet
  - CH Colmar, Colmar
  - CH Dieppe, Dieppe
  - CHU Dijon, Dijon
  - CH Sud Essonnes, Étampes
  - APHP, Garches
  - CHU Grenoble, Grenoble
  - CH Gueret, Guéret
  - CHU La Réunion, La Réunion
  - CHD Vendée, La Roche-sur-Yon
  - GH La Rochelle Ré Aunis, La Rochelle
  - CH Lens, Lens
  - GH de l'Institut Catholique de Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CH Meaux, Meaux
  - CH Melun, Melun
  - CHU Nantes, Nantes
  - CH Niort, Niort
  - CHU Nîmes, Nîmes
  - CHR Orleans, Orléans
  - APHP Cochin, Paris
  - APHP Saint Louis, Paris
  - Hôpital Paris Saint Joseph, Paris
  - CH Pau, Pau
  - CHU Poitiers, Poitiers
  - CH Pontoise, Pontoise
  - CH Cornouaille, Quimper
  - CH Roanne, Roanne
  - CHU Rouen, Rouen
  - CH Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rozen TH, Mullane S, Kaufman M, Hsiao YF, Warrillow S, Bellomo R, Jones DA. Antecedents to cardiac arrests in a teaching hospital intensive care unit. Resuscitation. 2014 Mar;85(3):411-7. doi: 10.1016/j.resuscitation.2013.11.018. Epub 2013 Dec 8. PMID 24326274
- [Background] Knaus WA, Zimmerman JE, Wagner DP, Draper EA, Lawrence DE. APACHE-acute physiology and chronic health evaluation: a physiologically based classification system. Crit Care Med. 1981 Aug;9(8):591-7. doi: 10.1097/00003246-198108000-00008. PMID 7261642
- [Background] Synek VM. EEG abnormality grades and subdivisions of prognostic importance in traumatic and anoxic coma in adults. Clin Electroencephalogr. 1988 Jul;19(3):160-6. doi: 10.1177/155005948801900310. PMID 3416501
- [Background] Myrianthefs P, Kalafati M, Lemonidou C, Minasidou E, Evagelopoulou P, Karatzas S, Baltopoulos G. Efficacy of CPR in a general, adult ICU. Resuscitation. 2003 Apr;57(1):43-8. doi: 10.1016/s0300-9572(02)00432-x. PMID 12668298
- [Background] Lesieur O, Leloup M, Gonzalez F, Mamzer MF; EPILAT Study Group. Eligibility for organ donation following end-of-life decisions: a study performed in 43 French intensive care units. Intensive Care Med. 2014 Sep;40(9):1323-31. doi: 10.1007/s00134-014-3409-2. Epub 2014 Aug 5. PMID 25091789
- [Background] Lee HK, Lee H, No JM, Jeon YT, Hwang JW, Lim YJ, Park HP. Factors influencing outcome in patients with cardiac arrest in the ICU. Acta Anaesthesiol Scand. 2013 Jul;57(6):784-92. doi: 10.1111/aas.12117. Epub 2013 Mar 31. PMID 23550795
- [Background] Peterson MW, Geist LJ, Schwartz DA, Konicek S, Moseley PL. Outcome after cardiopulmonary resuscitation in a medical intensive care unit. Chest. 1991 Jul;100(1):168-74. doi: 10.1378/chest.100.1.168. PMID 2060338
- [Background] Enohumah KO, Moerer O, Kirmse C, Bahr J, Neumann P, Quintel M. Outcome of cardiopulmonary resuscitation in intensive care units in a university hospital. Resuscitation. 2006 Nov;71(2):161-70. doi: 10.1016/j.resuscitation.2006.03.013. Epub 2006 Sep 20. PMID 16989937
- [Background] Landry FJ, Parker JM, Phillips YY. Outcome of cardiopulmonary resuscitation in the intensive care setting. Arch Intern Med. 1992 Nov;152(11):2305-8. PMID 1444691
- [Background] Tian J, Kaufman DA, Zarich S, Chan PS, Ong P, Amoateng-Adjepong Y, Manthous CA; American Heart Association National Registry for Cardiopulmonary Resuscitation Investigators. Outcomes of critically ill patients who received cardiopulmonary resuscitation. Am J Respir Crit Care Med. 2010 Aug 15;182(4):501-6. doi: 10.1164/rccm.200910-1639OC. Epub 2010 Apr 22. PMID 20413625
- [Background] Kutsogiannis DJ, Bagshaw SM, Laing B, Brindley PG. Predictors of survival after cardiac or respiratory arrest in critical care units. CMAJ. 2011 Oct 4;183(14):1589-95. doi: 10.1503/cmaj.100034. Epub 2011 Aug 15. PMID 21844108
- [Background] Smith DL, Kim K, Cairns BA, Fakhry SM, Meyer AA. Prospective analysis of outcome after cardiopulmonary resuscitation in critically ill surgical patients. J Am Coll Surg. 1995 Apr;180(4):394-401. PMID 7719542
- [Background] Cummins RO, Chamberlain D, Hazinski MF, Nadkarni V, Kloeck W, Kramer E, Becker L, Robertson C, Koster R, Zaritsky A, Bossaert L, Ornato JP, Callanan V, Allen M, Steen P, Connolly B, Sanders A, Idris A, Cobbe S. Recommended guidelines for reviewing, reporting, and conducting research on in-hospital resuscitation: the in-hospital 'Utstein style'. American Heart Association. Circulation. 1997 Apr 15;95(8):2213-39. doi: 10.1161/01.cir.95.8.2213. No abstract available. PMID 9133537
- [Background] Langhelle A, Nolan J, Herlitz J, Castren M, Wenzel V, Soreide E, Engdahl J, Steen PA; 2003 Utstein Consensus Symposium. Recommended guidelines for reviewing, reporting, and conducting research on post-resuscitation care: the Utstein style. Resuscitation. 2005 Sep;66(3):271-83. doi: 10.1016/j.resuscitation.2005.06.005. PMID 16129543
- [Background] Gershengorn HB, Li G, Kramer A, Wunsch H. Survival and functional outcomes after cardiopulmonary resuscitation in the intensive care unit. J Crit Care. 2012 Aug;27(4):421.e9-17. doi: 10.1016/j.jcrc.2011.11.001. Epub 2012 Jan 9. PMID 22227081
- [Background] Skrifvars MB, Varghese B, Parr MJ. Survival and outcome prediction using the Apache III and the out-of-hospital cardiac arrest (OHCA) score in patients treated in the intensive care unit (ICU) following out-of-hospital, in-hospital or ICU cardiac arrest. Resuscitation. 2012 Jun;83(6):728-33. doi: 10.1016/j.resuscitation.2011.11.036. Epub 2012 Jan 25. PMID 22281225
- [Background] Efendijev I, Raj R, Reinikainen M, Hoppu S, Skrifvars MB. Temporal trends in cardiac arrest incidence and outcome in Finnish intensive care units from 2003 to 2013. Intensive Care Med. 2014 Dec;40(12):1853-61. doi: 10.1007/s00134-014-3509-z. Epub 2014 Nov 12. PMID 25387815
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Lesieur O, Leloup M, Gonzalez F, Mamzer MF; EPILAT study group. Withholding or withdrawal of treatment under French rules: a study performed in 43 intensive care units. Ann Intensive Care. 2015 Dec;5(1):56. doi: 10.1186/s13613-015-0056-x. Epub 2015 Jun 19. PMID 26092498
- [Result] Leloup M, Briatte I, Langlois A, Cariou A, Lesieur O; ACIR study group. Unexpected cardiac arrests occurring inside the ICU: outcomes of a French prospective multicenter study. Intensive Care Med. 2020 May;46(5):1005-1015. doi: 10.1007/s00134-020-05992-w. Epub 2020 Mar 9. PMID 32152653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31,399 patients were admitted to intensive care unit (ICU), 24,245 were discharged alive without in-ICU cardiac arrest, 6,477 died in the ICU with no cardiopulmonary resuscitation (CPR) attempt, 677 had cardiac arrest with CPR attempt.
Groups:
- Shockable Rhythms: Patients with documented shockable rhythms during cardiac arrest
- Non-shockable Rhythms: Patients with documented non-shockable rhythms during cardiac arrest
Period: Overall Study
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Started | 120 | 557
Completed | 36 | 89
Not Completed | 84 | 468
Not completed — Death | 84 | 466
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shockable Rhythms | Non-shockable Rhythms | Total
Number analyzed (Participants) | 120 | 557 | 677
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 71 [60 to 78] | 69 [60 to 78] | 69 [60 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 175 | 210
  Male | 85 | 382 | 467
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 120 | 557 | 677

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Unexpected Cardiac Arrest
Description: Number of patients with at least one cardiac arrest in intensive care with attempted cardiopulmonary resuscitation as a proportion of total admissions.
Time Frame: 1 year
Population: Screening of all inpatients in the ICU during the study period. Only in-ICU cardiac arrest with attempted CPR are included in the study
Measure: Count of Participants; unit: Participants
Groups:
- In-ICU Admissions: Patients admitted in 45 participating intensive care unit (ICU) over one year
Arm/Group | In-ICU Admissions
Number analyzed (Participants) | 31,399
Participants
  in-ICU cardiac arrest with attempted CPR | 677
  No attempted CPR | 30,722

2. Secondary Outcome: Number of Patients Per Reason for ICU Admission
Description: Number of patients admitted to ICU with either Medical (vs surgical) reason for admission, circulatory failure, respiratory failure, cardiac arrest, cardiac surgery
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  Medical (vs surgical) reason for admission | 100 | 487
  Circulatory failure | 37 | 210
  Respiratory failure | 22 | 149
  Cardiac arrest | 31 | 69
  Cardiac surgery | 2 | 20

3. Secondary Outcome: History, Comorbidities Before Unexpected Cardiac Arrest
Description: High blood pressure, Diabetes, Dyslipidemia, Tobacco, Ischemic heart disease, Heart disease from another cause, Malignancy, Alcohol, Renal disease, Respiratory disease, Cardiac arrest, Neurological disease, Liver disease
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  High blood pressure | 75 | 322
  Diabetes | 37 | 182
  Dyslipidemia | 47 | 156
  Tobacco | 37 | 164
  Ischemic heart disease | 52 | 137
  Heart disease from another cause | 35 | 106
  Malignancy | 18 | 153
  Alcohol | 18 | 105
  Renal disease | 18 | 105
  Respiratory disease | 15 | 103
  Cardiac arrest | 8 | 41
  Neurological disease | 7 | 31
  Liver disease | 5 | 18

4. Secondary Outcome: Mc Cabe Score Before Unexpected Cardiac Arrest
Description: 0- absence of underlying disease or non-life-threatening disease
  1. underlying life-threatening disease over a period of 5 years
  2. underlying disease estimated fatal within 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  McCabe 0 (no fatal disease) | 63 | 269
  McCabe 1 or 2 | 57 | 288

5. Secondary Outcome: Knaus Score Before Unexpected Cardiac Arrest
Description: A- No activity limitation B- Moderate restriction of activity (limited professional activities) C- Major activity restriction but not total D- Major activity restriction, bedridden condition, long-term hospitalization
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  Knaus A or B (no or moderate limitation) | 92 | 392
  Knaus C or D | 28 | 165

6. Secondary Outcome: Organ Failure Score Before Unexpected Cardiac Arrest
Description: sequential organ failure assessment (SOFA) sub-score ≥ 3
  * Respiratory failure: < 200 fraction of inspired oxygen inspired oxygen fraction (26.7 mmHg [kilopascal]) and mechanically ventilated,
  * Neurological impairment : Glasgow coma scale <10,
  * Circulatory failure: dopamine > 5 μg/kg/min OR epinephrine ≤ 0.1 μg/kg/min OR norepinephrine ≤ 0.1 μg/kg/min,
  * Hepatic failure: ≥ 6.0-11.9 mg/dl [102-204 μmol/L] Bilirubin,
  * Haematological failure: < 50 Platelets×103/μl,
  * Renal failure: ≥ 3.5-4.9 mg/dl [300-44 0μmol/L] (or < 500 ml/d) Creatinine
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  Respiratory failure | 42 | 195
  Neurological impairment | 48 | 177
  Circulatory failure | 68 | 269
  Hepatic failure | 26 | 168
  Haematological failure | 3 | 63
  Renal failure | 2 | 25

7. Secondary Outcome: Number of Participants With Unexpected Cardiac Arrest Etiologies
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  At least one cause ultimately identified | 91 | 445
  Hypoxia | 15 | 164
  Metabolic disorder | 30 | 92
  Hypovolemia | 11 | 83
  Attributed to the life-sustaining device(s) | 11 | 87
  Respiratory support | 1 | 39
  Circulatory assistance | 7 | 32
  Medications | 3 | 19

8. Secondary Outcome: Number of Patients With Resumption of Spontaneous Cardiac Activity After Cardiopulmonary Resuscitation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants
  return of spontaneous circulation ≥ 20 min | 97 | 381
  return of spontaneous circulation ≥ 24 h | 73 | 223

9. Secondary Outcome: Cerebral Performance Category Scale at Hospital Discharge
Description: Cerebral performance category score (CPC)
  1. Conscious without neurological deficit or minor deficit
  2. Conscious with moderate deficit
  3. Conscious with severe deficit
  4. Deep Coma or Vegetative State
  5. Deceased
Time Frame: at Hospital Discharge
Measure: Count of Participants; unit: Participants
Groups:
- Shockable Rhythms and Alive at Hospital Discharge: Patients with documented shockable rhythms during cardiac arrest and alive at hospital discharge
- Non-shockable Rhythms and Alive at Hospital Discharge: Patients with documented non-shockable rhythms during cardiac arrest and alive at hospital discharge
Arm/Group | Shockable Rhythms and Alive at Hospital Discharge | Non-shockable Rhythms and Alive at Hospital Discharge
Number analyzed (Participants) | 44 | 102
Participants
  CPC 1 or 2 | 43 | 92
  CPC 3 | 1 | 8
  CPC 4 | 0 | 2

10. Secondary Outcome: Cerebral Performance Category Scale at 6 Months
Description: as for outcome 9
Time Frame: at 6 months after inclusion (unexpected cardiac arrest)
Measure: Count of Participants; unit: Participants
Groups:
- Shockable Rhythms and Alive at 6-month Follow-up: Patients with documented shockable rhythms during cardiac arrest and alive at 6-month follow-up
- Non-shockable Rhythms and Alive at 6-month Follow-up: Patients with documented non-shockable rhythms during cardiac arrest and alive at 6-month follow-up
Arm/Group | Shockable Rhythms and Alive at 6-month Follow-up | Non-shockable Rhythms and Alive at 6-month Follow-up
Number analyzed (Participants) | 36 | 89
Participants
  CPC 1 or 2 | 36 | 82
  CPC 3 | 0 | 6
  CPC 4 | 0 | 1

11. Secondary Outcome: Number of Patients With Unexpected Cardiac Arrest, Resuscitated Despite Previous Decision Not to Resuscitate
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Shockable Rhythms | Non-shockable Rhythms
Number analyzed (Participants) | 120 | 557
Participants | 2 | 11

ADVERSE EVENTS:
Time Frame: 6-month follow up
Arm/Group | In-ICU Admissions
All-Cause Mortality (participants affected / at risk) | 550/677
Serious Adverse Events (participants affected / at risk) | 7/677
Other Adverse Events (participants affected / at risk) | 118/677
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-ICU Admissions (N=677)
Conscious with severe deficit (Nervous system disorders) | 7 (20)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-ICU Admissions (N=677)
Conscious without neurological deficit, minor or moderate deficit (Nervous system disorders) | 118 (143)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03021564/Prot_SAP_ICF_000.pdf